CLINICAL TRIAL: NCT07328633
Title: Effect of Pre-habilitation Combined With Enhanced Recovery After Surgery (ERAS) Versus ERAS Perioperative Management on Clinical Outcomes of Laparoscopic (Robotic) Gastrectomy in Patients With Gastric Cancer Receiving Neoadjuvant Chemotherapy: A Single-center Randomized Controlled Trial
Brief Title: Prehabilitation Plus ERAS in Gastric Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Principal Investigator, Zhou Yanbing, chief physician, The Affiliated Hospital of Qingdao University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QYFYEC2025-08
Record Dates: First submitted 2025-09-19; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Gastric Cancer (GC)
Keywords: Gastric Cancer; Neoadjuvant Chemotherapy; Laparoscopic Gastrectomy; Robotic Surgery; Pre-habilitation; Enhanced Recovery After Surgery (ERAS)
MeSH Terms: conditions — Stomach Neoplasms | interventions — Enhanced Recovery After Surgery; Clinical Protocols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-habilitation + ERAS (Experimental): Participants will undergo a 4-week pre-habilitation program including exercise, nutrition, and psychological support, followed by Enhanced Recovery After Surgery (ERAS) protocols.
  Interventions: Behavioral: Pre-habilitation Program; Procedure: Enhanced Recovery After Surgery (ERAS) Protocol
- ERAS Only (Active Comparator): Participants will receive standard Enhanced Recovery After Surgery (ERAS) protocols without the pre-habilitation program.
  Interventions: Procedure: Enhanced Recovery After Surgery (ERAS) Protocol

INTERVENTIONS:
Behavioral: Pre-habilitation Program — A 4-week pre-habilitation program including exercise, nutrition, and psychological support aimed at improving physical and mental readiness for surgery.
  Arms: Pre-habilitation + ERAS
Procedure: Enhanced Recovery After Surgery (ERAS) Protocol — Standard protocols for Enhanced Recovery After Surgery aimed at reducing postoperative complications and accelerating recovery.

SUMMARY:
This study aims to evaluate the impact of pre-habilitation combined with Enhanced Recovery After Surgery (ERAS) versus ERAS perioperative management alone on clinical outcomes in patients with gastric cancer undergoing neoadjuvant chemotherapy and laparoscopic (robotic) gastrectomy. The study is a single-center, randomized controlled trial involving patients aged 18-75 years. Participants will be randomly assigned to either a pre-habilitation program plus ERAS or ERAS alone. The primary outcome is the incidence of postoperative complications within 30 days. Secondary outcomes include pathological data, surgical outcomes, patient-reported outcomes, and long-term survival rates.

DETAILED DESCRIPTION:
The study is designed as a prospective, single-center, randomized, open-label, controlled clinical trial to compare the effects of pre-habilitation combined with ERAS versus ERAS alone in patients undergoing laparoscopic (robotic) gastrectomy after neoadjuvant chemotherapy for gastric cancer. The study will enroll patients aged 18-75 years who are scheduled for laparoscopic (robotic) gastrectomy following neoadjuvant chemotherapy. Participants will be randomly assigned in a 1:1 ratio to either the pre-habilitation plus ERAS group or the ERAS group. The pre-habilitation program will include a 4-week intervention involving exercise, nutrition, and psychological support prior to surgery. The primary endpoint is the incidence of postoperative complications within 30 days, assessed using the Clavien-Dindo classification. Secondary endpoints include pathological characteristics, surgical outcomes, patient-reported outcomes, and long-term survival rates. Data will be collected from patient records and follow-up visits. Statistical analysis will be performed using SPSS 26.0 or later versions, with significance level set at α=0.05.

ELIGIBILITY:
Inclusion Criteria:

* Age:18-75 years
* ECOG:0-2
* ASA:I-III
* Histologically confirmed gastric adenocarcinoma (cT3-4aN+M0)
* Fit for radical surgery after MDT
* Negative pregnancy test within one month
* Non-pregnant or non-lactating

Exclusion Criteria:

* Severe cardiac (LVEF<30% or NYHA IV)
* Severe hepatic or renal dysfunction (Child-Pugh ≥10; CrCl<25 ml/min)
* Recent cerebrovascular events
* Concomitant tumors requiring surgery
* Emergency surgery for tumor complications,
* Severe infections

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2024-12-05 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Postoperative Complications | Postoperative 30-day
  The primary outcome measure is the incidence of postoperative complications within 30 days after surgery, assessed using the Clavien-Dindo classification system(CDC ≥ II).

SECONDARY OUTCOMES:
Operation time | Intra-operative
  Time from skin incision to skin closure. Unit: minutes.
Estimated blood loss | Intra-operative
  Total volume of intra-operative blood loss. Unit: mL.
Pathological ypT stage | At pathology review (within 2 week after surgery)
  Tumour infiltration depth in the resection specimen according to AJCC 8th edition.
  Unit: n (%) - categories T0, T1, T2, T3, T4.
Pathological ypN stage | At pathology review (within 2 week after surgery)
  Number of metastatic lymph nodes in the resection specimen. Unit: n (%) - categories N0, N1, N2, N3.
AJCC pathological TNM stage | At pathology review (within 2 week after surgery)
  Combined pathological stage. Unit: n (%) - stages I, II, III.
Tumour regression grade (TRG) | At pathology review (within 2 week after surgery)
  Degree of tumour response to neoadjuvant therapy according to Mandard criteria. Unit: n (%) - grades 0, 1, 2, 3.
Time to first flatus | Post-operative period (up to 30 days)
  Interval from end of surgery to first rectal gas passage. Unit: days.
Time to first liquid diet | Post-operative period (up to 30 days)
  Interval from end of surgery to first tolerated liquid intake. Unit: days.
Post-operative hospital stay | Post-operative period.
  Interval from surgery to hospital discharge. Unit: days.
Serum albumin level | Post-operative day 1,3,5.
  Serum albumin measured post-operatively. Unit: g/L.
Tumour differentiation | At pathology review (within 2 week after surgery)
  Histological grade of the tumour. Unit: n (%) - well / moderate / poor.

OTHER OUTCOMES:
Sex distribution | Baseline (day of enrollment)
  Biological sex at enrollment Unit: n (%) - Male, Female
Height | Baseline (day of enrollment)
  Body height measured without shoes Unit: cm
Weight | Baseline (day of enrollment)
  Body weight measured in light indoor clothing Unit: kg
ECOG performance status | Baseline (day of enrollment)
  Eastern Cooperative Oncology Group performance score Unit: n (%) - scores 0, 1, 2
Nutritional risk score (NRS 2002) | Baseline (day of enrollment)
  Nutritional Risk Screening 2002 total score Unit: n (%) - <3 vs ≥3
ASA physical status classification | Baseline (day of enrollment)
  American Society of Anesthesiologists classification Unit: n (%) - classes 1, 2, 3
Tumor diameter | Baseline (after neoadjuvant therapy, before surgery)
  Maximum diameter of the primary tumor on pre-operative imaging Unit: cm
Clinical T stage | Baseline (after neoadjuvant therapy, before surgery)
  Clinical T category per AJCC 8th edition Unit: n (%) - cT2, cT3, cT4
Clinical N stage | Baseline (after neoadjuvant therapy, before surgery)
  Clinical N category per AJCC 8th edition Unit: n (%) - cN0, cN1, cN2, cN3
Six-minute walk test distance | Baseline (after neoadjuvant therapy, before surgery)
  Distance walked in 6 minutes on indoor flat track Unit: meters
Hospital Anxiety and Depression Scale (HADS) | From the end of neoadjuvant therapy to the day before surgery, assessed up to 42 days.
  Anxiety and depression symptoms assessed with the 14-item HADS questionnaire; total score 0-21, higher scores indicate greater symptom severity.
  Unit: score (0-21)
Health-related quality of life (EORTC QLQ-C30) | From the end of neoadjuvant therapy to the day before surgery, assessed up to 42 days.
  Assessed with the 30-item EORTC QLQ-C30 questionnaire; 15 domains (5 functional, 9 symptom/single-item, 1 global QoL). Raw scores are linearly transformed to 0-100 standard scores. Higher functional/global scores = better QoL; higher symptom scores = worse symptoms.
  Unit: score (0-100)

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) including baseline demographics, intervention details, and all primary/secondary outcomes will be shared. No participant identifiers will be included.
Supporting Information: Study Protocol
Time Frame: Start date:Main results publication date. End date:5 years after publication.
Access Criteria: Data will be available to qualified researchers upon reasonable request. Requests should be sent to 17866805578@163.com with a brief research proposal. A data-sharing agreement is required. Data will be provided in CSV format within 3 months of request approval.
URL: https://pan.baidu.com/s/1T1f9IojYhtnVAkT8gLZryg

REFERENCES:
- [Result] Ajani JA, Bentrem DJ, Besh S, D'Amico TA, Das P, Denlinger C, Fakih MG, Fuchs CS, Gerdes H, Glasgow RE, Hayman JA, Hofstetter WL, Ilson DH, Keswani RN, Kleinberg LR, Korn WM, Lockhart AC, Meredith K, Mulcahy MF, Orringer MB, Posey JA, Sasson AR, Scott WJ, Strong VE, Varghese TK Jr, Warren G, Washington MK, Willett C, Wright CD, McMillian NR, Sundar H; National Comprehensive Cancer Network. Gastric cancer, version 2.2013: featured updates to the NCCN Guidelines. J Natl Compr Canc Netw. 2013 May 1;11(5):531-46. doi: 10.6004/jnccn.2013.0070. PMID 23667204
- [Result] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Result] Xing J, Wang Y, Shan F, Li S, Jia Y, Ying X, Zhang Y, Li Z, Ji J. Comparison of totally laparoscopic and laparoscopic assisted gastrectomy after neoadjuvant chemotherapy in locally advanced gastric cancer. Eur J Surg Oncol. 2021 Aug;47(8):2023-2030. doi: 10.1016/j.ejso.2021.02.002. Epub 2021 Feb 6. PMID 33663942
- [Result] Zhong H, Liu X, Tian Y, Cao S, Li Z, Liu G, Sun Y, Zhang X, Han Z, Meng C, Jia Z, Wang Q, Zhou Y. Comparison of short- and long-term outcomes between laparoscopic and open gastrectomy for locally advanced gastric cancer following neoadjuvant chemotherapy: a propensity score matching analysis. Surg Endosc. 2023 Aug;37(8):5902-5915. doi: 10.1007/s00464-023-10052-7. Epub 2023 Apr 18. PMID 37072637
- [Result] Liu G, Cao S, Liu X, Tian Y, Li Z, Sun Y, Zhong H, Wang K, Zhou Y. Short- and long-term outcomes following perioperative ERAS management in patients undergoing minimally invasive radical gastrectomy after neoadjuvant chemotherapy: A single-center retrospective propensity score matching study. Eur J Surg Oncol. 2025 Jan;51(1):109459. doi: 10.1016/j.ejso.2024.109459. Epub 2024 Nov 15. PMID 39566200

DOCUMENTS (2):
  • Study Protocol (2024-07-27): https://cdn.clinicaltrials.gov/large-docs/33/NCT07328633/Prot_000.pdf
  • Informed Consent Form (2024-07-27): https://cdn.clinicaltrials.gov/large-docs/33/NCT07328633/ICF_001.pdf